CLINICAL TRIAL: NCT05721456
Title: A Phase 3, Randomized, Partially-Blind, Clinical Trial to Evaluate the Non-Inferiority of a 12-Valent Pneumococcal Conjugate Vaccine in Healthy Children in Brazil, Compared to 10- and 13-Valent Pneumococcal Conjugate Vaccines
Brief Title: Evaluation of the Non-Inferiority of a 12-Valent Pneumococcal Conjugate Vaccine in Healthy Children in Brazil.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maria de Lourdes de Sousa Maia, MD (Other)
Responsible Party: Sponsor-Investigator, Maria de Lourdes de Sousa Maia, MD, Sponsor, The Immunobiological Technology Institute (Bio-Manguinhos) / Oswaldo Cruz Foundation (Fiocruz)
Organization: The Immunobiological Technology Institute (Bio-Manguinhos) / Oswaldo Cruz Foundation (Fiocruz) (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Protocol ASCLIN 002/2022
Record Dates: First submitted 2022-11-23; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-01

CONDITIONS: Pneumococcal Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PCV10 (Synflorix®) (Active Comparator)
  Interventions: Biological: 12-Valent Pneumococcal Conjugate Vaccine
- PCV13 (Prevenar13®) (Active Comparator)
  Interventions: Biological: 12-Valent Pneumococcal Conjugate Vaccine
- 12-Valent Pneumococcal Conjugate Vaccine (Experimental)
  Interventions: Biological: 12-Valent Pneumococcal Conjugate Vaccine

INTERVENTIONS:
Biological: 12-Valent Pneumococcal Conjugate Vaccine — PCV12 group 1: 550 subjects receiving the 12-valent pneumococcal polysaccharide conjugate vaccine (12Pn-PD-DiT-CRM), defined as PCV12 in this protocol
  Other Names: PCV12

SUMMARY:
The purpose of this phase III study is to demonstrate immunologic non-inferiority in terms of proportion of individuals with antibody concentration ≥0.2 µg/mL (by modified 22F-inhibition enzyme-linked immunosorbent assay, ELISA) or in terms of ELISA geometric mean concentrations (GMC) of serotype-specific IgG, of 12-valent pneumococcal polysaccharide conjugate vaccine (12Pn-PD-DiT-CRM, hereby indicated as PCV12), containing the serotypes 1, 4, 5, 6B, 7F, 9V, 14, and 23F conjugated with non-typeable Haemophilus influenzae protein D, 19F conjugated with TD, 18C conjugated with TT, and 6A and 19A conjugated with CRM197, and to assess its safety in the population of infants vaccinated from 2 months of age with a primary regimen of 2 or 3 doses plus a booster administered at one year of life.

DETAILED DESCRIPTION:
The purpose of this phase III study is to demonstrate immunologic non-inferiority in terms of proportion of individuals with antibody concentration ≥0.2 µg/mL (by modified 22F-inhibition enzyme-linked immunosorbent assay, ELISA) or in terms of ELISA geometric mean concentrations (GMC) of serotype-specific IgG, of 12-valent pneumococcal polysaccharide conjugate vaccine (12Pn-PD-DiT-CRM, hereby indicated as PCV12), containing the serotypes 1, 4, 5, 6B, 7F, 9V, 14, and 23F conjugated with non-typeable Haemophilus influenzae protein D, 19F conjugated with TD, 18C conjugated with TT, and 6A and 19A conjugated with CRM197, and to assess its safety in the population of infants vaccinated from 2 months of age with a primary regimen of 2 or 3 doses plus a booster administered at one year of life. Hence, this study will provide non-inferiority evidence for possible approval of a new pneumococcal vaccine in Brazil and its eventual inclusion in the national immunization program (PNI). PCV12 will be produced in national facilities, after transfer of technology to Bio-Manguinhos/Fiocruz, thus ensuring continuous provision to the public healthcare system (SUS).

This study is designed to demonstrate the immunologic non-inferiority of the PCV12 for each one of the 12 vaccine pneumococcal serotypes, when compared to the licensed vaccines GSK Synflorix® (PCV10) and Pfizer's/Wyeth's Prevenar 13® (PCV13). PCV10 will be used for the comparison of the immune response to the 10 common serotypes. PCV13 or the least immunogenic serotype of PCV10 will be used for the comparison of the immune response to the two additional pneumococcal serotypes 19A and/or 6A conjugated to CRM197.

The non-inferiority of PCV12 will be evaluated in the two schedules recommended in Brazil, the 2+1 scheme (followed by PNI) or the 3+1 scheme (the reference schedule when evaluating new vaccines).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, 6-12 weeks of age, inclusive, at the time of the first vaccination.
2. Healthy subjects as established by medical history and clinical examination before entering into the study.
3. Subjects who the investigator believes that parent(s)/ Legally Acceptable Representative(s) [LAR(s)] can and will comply with the requirements of the protocol, including:

   1. willing to provide name, address, and telephone number for contact if necessary (e.g., in case of missing a scheduled visit)
   2. available for follow-up throughout the study period
   3. capable to complete the forms for registration of signs and symptoms at home.
4. Parent(s)/LAR(s) are able to understand and sign the informed consent form.

Exclusion Criteria:

1. Preterm infants (gestation <36 weeks) or with low birth weight (<2000g).
2. Use of any investigational or non-registered product other than the study vaccines and allowed co-administered vaccines as outlined in section 3.4.9. during the entire study period. Any other vaccine administration must be discussed and approved by the medical monitor.
3. Medical history of culture- or PCR-confirmed invasive disease caused by S. pneumoniae.
4. Coagulation problems.
5. Chronic administration (more than 14 days in total) of corticosteroids, immunosuppressants or other immune-modifying drugs (except palivizumab) since birth or planned use during the study.
6. Administration of immunoglobulins and/or blood products since birth or planned use during the study period.
7. Participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
8. Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
9. History of any reaction or hypersensitivity likely to be exacerbated by any component of the study vaccine.
10. Major congenital defects or serious chronic illness.
11. History of any seizures or any neurological disease
12. Acute disease and/or fever (axillary temperature ≥38ºC) at the time of enrolment.
13. Previous vaccination with any pneumococcal vaccine.
14. Infants born of woman who received any pneumococcal vaccine during pregnancy.

Ages: 2 Months to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2400 (Estimated)
Dates: Start 2023-08-28 (Estimated); Primary Completion 2024-04-28 (Estimated); Study Completion 2025-01-28 (Estimated)

PRIMARY OUTCOMES:
The immunological non-inferiority of pneumococcal vaccine 12 in relation to pneumococcal vaccine 10 and 13. | 5 months
  Proportion of subjects with serotype-specific pneumococcal IgG antibody concentration ≥0.20 µg/mL after primary vaccination.Geometric mean concentrations of serotype-specific pneumococcal IgG antibody after primary vaccination.

SECONDARY OUTCOMES:
Functional Antibody Response | 17 months
  Opsonophagocytic activity (OPA) for antibodies against each of the pneumococcal serotypes 1, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F will be measured by a killing-assay using a HL 60 cell line (37) or using a multiplex assay. The results will be presented as the dilution of serum (opsonic titer) able to sustain 50% killing of live pneumococci under the assay conditions, as geometric mean titers (GMTs). The defined cut-off of the assay is an opsonic titer of 8, and percentage of children with titers ≥8 will also be presented for each serotype.
  Paired samples of the same individual will also be tested, however, without breaking the blinding relative to the time of collection (pre or post vaccination) and the type of vaccine received (experimental or comparators).
Immunogenicity after booster | 17 months
  Pneumococcal serotype specific total IgG antibodies (antibodies to 1, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) will each be measured by 22F-inhibition ELISA). The antibody concentration will be determined by logistic log comparison of the ELISA curves with a standard reference serum 89-SF or SP007 available from the US Food and Drug Administration for which concentration of IgG to the 12 serotypes are known in μg/mL . The cut-off of the assay is 0.05 μg/mL. For each group, immune responses to each serotype will be expressed as antibody GMCs and the percentage of children with IgG concentrations ≥0.2 μg/mL that is equivalent to concentrations of ≥0.35 μg/mL measured by the non-22F ELISA, of the World Health Organization reference laboratory.
  Samples of the same individual will be tested in a paired manner but without breaking the blinding relative to the time of collection (pre or post vaccination) and the type of vaccine received (experimental or comparators).
Safety and reactogenicity vaccination and booster vaccination. | 18 months
  Proportion of subjects with any and Grade 3 solicited local adverse event (AE) within 7 days after each vaccination dose.
  • Proportion of subjects with any and Grade 3 solicited systemic AE, within 7 days after each vaccination dose.
  Solicited systemic AEs include drowsiness, irritability/agitation, loss of appetite and fever (axillary temperature ≥ 38°C).
  • Proportion of subjects with any solicited or unsolicited AEs after each vaccination dose.
  on.
  * Proportion of subjects with any serious adverse event (SAE) after last dose of primary vaccination.
  * Proportion of subjects with any SAE after booster vaccination.
Immunogenicity, safety and reactogenicity co-administered vaccines | 17 months
  Due to the restriction of collecting larger volumes of blood in young children, this analysis will be restricted to a subsample of 120 study subjects (60 per schedule, 20:20:20 per vaccination group), randomly selected and without breaking study blinding.The evaluation of antitetanic and anti-diphteric antibodies, and of IgG specific for purified capsular polysaccharides from Neisseria meningitidis serogroup C, present in the volunteer sera will be performed in Bio-Manguinhos/Fiocruz, assessed by the immunoenzymatic technique (ELISA) and expressed in international units per milliliter of serum (IU/mL). Paired samples of the same individual will also be tested, however, without breaking the blinding relative to the time of collection (pre or post vaccination) and the type of vaccine received (experimental or comparators).